CLINICAL TRIAL: NCT00241709
Title: Case-Control Association Studies and Genetic Confounding
Brief Title: Optimal Approach for Analysis of Case-Control Genetic Association Studies
Acronym: GALA 1
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1309; R01HL078885 (NIH)
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Retrospective genetic analysis of DNA; samples collected between 1998-2001
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the effectiveness of approaches to correct for the effects of population stratification on case-control genetic association studies.

DETAILED DESCRIPTION:
BACKGROUND:

In racially admixed populations, genetic associations may be confounded by population stratification. To control for population stratification, statistical methods that use marker genotype data to infer population structure have been proposed as an alternative to family-based tests of association. However, there are limited empirical data on how these methods perform in real populations. This study will use well characterized populations of Mexican and Puerto Rican asthmatics, their parents, and control subjects recruited from the same sites to examine the effectiveness of approaches to correct for the effects of population stratification on case-control genetic association studies.

DESIGN NARRATIVE:

This study has three specific aims: 1) To test and compare methods of detecting and correcting for population stratification, the study will genotype a total of 100 ancestral informative markers (AIMs) for 400 asthma cases and an equal number of control subjects. These AIMs will then be used with three statistical methods developed to detect and correct for population stratification. The number and characteristics of markers required to correct false positive associations between AIMs, asthma, and asthma quantitative traits will be evaluated and compared; 2) To compare the power of genomically adjusted case-control studies to the Transmission Disequilibrium Test (TDT). An allele from each of the 100 AIMs will be considered as a risk factor for a simulated "phenotype." The association between phenotypes and each AIM will be tested with the TDT and with a case-control analysis after adjustment for stratification to compare the false negative rates for these study designs. 3) To use the results from aim 1 and 2 to define an optimal approach for analysis and interpretation of case-control association studies in these populations and apply this approach to analyze the association between asthma and a series of candidate genes. The results of these studies should provide important insights into optimal methods to control for population stratification in case-control association studies, thereby facilitating the inclusion of admixed populations in future genetic studies of complex diseases such as asthma.

ELIGIBILITY:
No eligibility criteria; this study will be using existing blood samples of Mexican and Puerto Rican asthmatics, their parents, and control participants who were recruited prior to the study.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Family-based cross sectional analysis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2005-08; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Gonzalez Burchard, MD, Principal Investigator — University of California School of Medicine, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States